CLINICAL TRIAL: NCT00899652
Title: The Molecular Epidemiology of de Novo and Treatment Related 11q23 Leukemia in the Young
Brief Title: DNA Analysis of Bone Marrow and Blood Samples From Young Patients With Acute Myeloid Leukemia or Acute Lymphoblastic Leukemia
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: B945; CCG-B945 (Other: Children's Cancer Group); CDR0000538662 (Other: Clinical Trials.gov); COG-B945 (Other: Children's Oncology Group)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Leukemia
Keywords: childhood acute myelomonocytic leukemia (M4); childhood acute monocytic leukemia (M5b); childhood acute monoblastic leukemia (M5a); secondary acute myeloid leukemia; untreated childhood acute lymphoblastic leukemia; untreated childhood acute myeloid leukemia and other myeloid malignancies; recurrent childhood acute lymphoblastic leukemia; recurrent childhood acute myeloid leukemia
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Blotting, Southern; Cytogenetic Analysis; Gene Rearrangement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — marrow, blood, pheresis bag
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All Patients: Completion of Telephone Study Entry Form, Additional On Study Form, and Specimen Transmittal Form.
  Interventions: Genetic: Southern blotting; Genetic: chromosomal translocation analysis; Genetic: cytogenetic analysis; Genetic: gene rearrangement analysis; Genetic: mutation analysis

INTERVENTIONS:
Genetic: Southern blotting
Genetic: chromosomal translocation analysis
Genetic: cytogenetic analysis
Genetic: gene rearrangement analysis
Genetic: mutation analysis

SUMMARY:
RATIONALE: Studying samples of bone marrow and blood from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This laboratory study is looking at DNA in bone marrow and blood samples from young patients with acute myeloid leukemia or acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Characterize the clinical, morphologic, immunologic, cytogenetic, and molecular heterogeneity of acute lymphoblastic leukemia or acute myeloid leukemia (AML) in infants and monoblastic variants of AML in young patients.
* Characterize the clinical, morphologic, immunologic, cytogenetic, and molecular heterogeneity of secondary AML in young patients.
* Compare secondary AML vs de novo AML at the level of Southern blot, breakpoint sequence, and DNA topoisomerase II cleavage sites.

OUTLINE: This is a multicenter study.

Bone marrow or blood are collected and analyzed by Southern blot for chromosome 11q23 breakpoints and translocations. Samples from patients with secondary acute myeloid leukemia are also examined for MLL gene rearrangements.

PROJECTED ACCRUAL: A total of 250 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of leukemia meeting 1 of the following criteria:

  * Acute lymphoblastic leukemia OR acute myeloid leukemia (AML) (< 1 year of age at diagnosis)
  * M4 OR M5 AML (< 5 years of age at diagnosis)
  * Secondary leukemia (< 21 years of age at diagnosis)
* Bone marrow sample, peripheral blood (WBC > 10,000/mm³ and 20% peripheral blasts), or pheresis bag available

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 149 (Actual)
Dates: Start 1997-01; Primary Completion 2005-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Clinical, morphologic, immunologic, cytogenetic, and molecular characteristics of acute lymphoblastic leukemia and de novo and secondary acute myeloid leukemia (AML)
Comparison of secondary AML vs de novo AML at the level of Southern blot, breakpoint sequence, and DNA topoisomerase II cleavage sites

CONTACTS AND LOCATIONS:
Overall Officials: Beverly J. Lange, MD, Study Chair — Children's Hospital of Philadelphia; Carolyn A. Felix, MD — Children's Hospital of Philadelphia